CLINICAL TRIAL: NCT00775541
Title: Hyperglycemia and Oxidative Stress in the Human Brain With Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient dose for MRI scanning
Sponsor: In-Young Choi, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, In-Young Choi, Ph.D., Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 11066; GCRC CReff 0082
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2012-06-18 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin C (Experimental): 2 gms vitamin C
  Interventions: Dietary Supplement: Vitamin C

INTERVENTIONS:
Dietary Supplement: Vitamin C — One IV infusion of 2 gm vitamin C

SUMMARY:
The purpose of this study is to use an MRI exam to measure the concentrations of glutathione (GSH) and Vitamin C (Asc) in the brains of normal healthy persons and type 2 diabetic persons. The study will look at the relationship between chronic hyperglycemia and the levels of these naturally occurring chemicals in the brain.

DETAILED DESCRIPTION:
Cerebral GSH and Asc concentrations are modulated by increased oxidative stress induced by hyperglycemia in diabetes and reflect changes in the cerebral antioxidant defense system. Inhibition of cellular uptake of Asc by hyperglycemia further hampers maintaining adequate antioxidant capacities. Reduced concentrations of these antioxidants might serve as good indicators of increased susceptibility to oxidative damage, impaired cellular uptake or the antioxidant, and further, as sensitive in vivo biomarkers to assess early manifestations or progression of diabetic complications and the efficacy of the antioxidant therapy in the human brain. Specific aims (1) to determine cerebral concentrations of GSH and Asc in the living brain of healthy controls and type 2 diabetic patients; (2) to quantify the effect of chronic hyperglycemia on cellular uptake of Asc across the blood-brain barrier.

ELIGIBILITY:
Inclusion Criteria:

* Good health except for having type 2 diabetes
* Being treated with diet, insulin, or oral hyperglycemic agents
* Male or non pregnant female
* Non-smoker
* HbA1c 8 or above
* Able to provide informed consent

Exclusion Criteria:

* Presence of mental illness
* Co-existing chronic inflammatory condition or neurological disease or diseases associated with abnormal glutathione metabolism
* BMI over 35
* Smoker

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2007-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
MRI, mRS, urine and blood samples | before and after IV infusion, 6 hours

SECONDARY OUTCOMES:
7 day food and DHQ food questionnaire | 7 days prior to MRI and vitamin C infusion

CONTACTS AND LOCATIONS:
Overall Officials: In-Young Choi, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States